CLINICAL TRIAL: NCT04083339
Title: Aldose Reductase Inhibition for Stabilization of Exercise Capacity in Heart Failure (ARISE-HF): A Multicenter, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of AT-001 in Patients With Diabetic Cardiomyopathy
Brief Title: Safety and Efficacy of AT-001 in Patients With Diabetic Cardiomyopathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-001-2001
Record Dates: First submitted 2019-08-23; First posted 2019-09-10 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Cardiomyopathies
Keywords: Type 2 Diabetes; Aldose Reductase Inhibitor; Stage B Heart Failure; Stage C Heart Failure; Cardiopulmonary Exercise Test
MeSH Terms: conditions — Diabetic Cardiomyopathies; Diabetes Mellitus, Type 2 | interventions — caficrestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AT-001 High dose (Experimental): The total daily doses will be of 3g. The dose selection and the frequency of dosing was based on the results of the phase 1/2 study demonstrating that 3g/day of AT-001 is capable of producing the maximum inhibition of the production of sorbitol (a pharmacodynamic biomarker of biological activity).
  Interventions: Drug: AT-001
- AT-001 Low Dose (Experimental): The total daily doses will be of 2g. The dose selection and the frequency of dosing was based on the results of the phase 1/2 study demonstrating that 2g/day of AT-001 is capable of producing a sufficient inhibition of the production of sorbitol (a pharmacodynamic biomarker of biological activity).
  Interventions: Drug: AT-001
- Placebo Comparator (Placebo Comparator): Placebo capsules will be used as comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AT-001 — AT-001 will be administered as 3 capsules twice daily, before breakfast and before dinner.
  At present AT001 is the sole name for the active substance. No INN/genetic name is available to date
  Arms: AT-001 High dose; AT-001 Low Dose
Drug: Placebo — Matching placebo will be administered as 3 capsules twice daily, before breakfast and before dinner
  Arms: Placebo Comparator

SUMMARY:
This is a multicenter, randomized, placebo-controlled, 2-part study to evaluate the safety and efficacy of AT-001 in adult patients (N=675) with Diabetic Cardiomyopathy at high risk of progression to overt heart failure.

DETAILED DESCRIPTION:
The study consists of two consecutive parts: Part A and Part B. Part A will evaluate the safety and efficacy of two doses of AT-001 vs placebo. The primary objective of Part A is to demonstrate that AT-001 improves or prevents the decline of functional capacity in patients with Diabetic Cardiomyopathy. Part B is an extension of at least 12 months that will evaluate the safety and efficacy of chronic administration of AT-001 vs placebo in the same patients who had previously been evaluated in Part A. Assessments in Part B will include safety endpoints and exploratory clinical efficacy endpoints, i.e. death and hospitalization due to a cardiac event.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Diabetic cardiomyopathy
* Peak VO2 < 75% of predicted normal value based on age and gender

Exclusion Criteria:

* Prior diagnosis or signs/symptoms of overt/symptomatic heart failure / stage C heart failure
* Prior echocardiogrphic measurement of ejection fraction (EF) < 40%
* Prior acute coronary syndrome (ACS), coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), coronary artery disease (CAD) or stroke
* Severe or moderate cardiac valve disease requiring intervention
* Clinically significant arrhythmia
* Prior diagnosis of congenital, infective, toxic, infiltrative, post-partum, or hypertrophic cardiomyopathy
* Blood pressure > 140 mmHg (systolic) or > 90 mmHg (diastolic) at screening
* HbA1c >8.5% at screening
* Severe disease that would impact the performance of a cardio-pulmonary exercise test

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 during cardio-pulmonary exercise test (CPET); | 15 months after randomization]
  Changes in Peak VO2 during cardio-pulmonary exercise test (CPET) from baseline to approximately Month 15 (15-18 months). A CPET may be repeated at approximately Month 27 (27-30 months).

SECONDARY OUTCOMES:
Progression to overt heart failure (Stage C Heart Failure) | 27 months after randomization
  Defined by the occurrence of one of the following events: cardiovascular death, hospitalization for heart failure, urgent heart failure visit, new diagnosis of heart failure
Changes in NT-proBNP | 27 months after randomization
  Changes in NT-proBNP may reflect worsening of cardiomyopathy over time
Changes in the modified Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 27 months after randomization
  Changes in the modified KCCQ may reflect deterioration of clinical status over time

OTHER OUTCOMES:
Worsening of diabetic cardiomyopathy | 15 and 27 months after randomization
  Defined by either ≥ 20% increase in NT-proBNP or ≥ 5 point decrease in the mKCCQ score
Changes in echocardiographic parameters | 27 months after randomization
  Changes assessed on cardiac ultra-sound from baseline

CONTACTS AND LOCATIONS:
Overall Officials: James L Januzzi, MD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (79):
- United States (28):
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - University of California, San Diego (UCSD), La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - University of California - Irvine Medical Center, Orange, California
  - Metabolic Institute of America, Tarzana, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - UnityPoint Health - Methodist Hospital, Peoria, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Universty of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Heart and Vascular Cardiology, St Louis, Missouri
  - Chear Center LLC, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Remington Davis, Inc., Columbus, Ohio
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Mountain View Clinical Research - Greer, Greer, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Juno Research, LLC - Northwest Site, Houston, Texas
  - Juno Research, LLC - Southwest Houston Site, Houston, Texas
  - FMC Science, Lampasas, Texas
- Australia (7):
  - Prince Charles Hospital, Chermside, Queensland
  - CORE Research Group Pty. Ltd., Milton, Queensland
  - AusTrials, Taringa, Queensland
  - University of Tasmania at Hobart, Hobart, Tasmania
  - Barwon Health-University Hospital Geelong, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
- Canada (9):
  - C-Endo - Endocrinology Centre, Calgary, Alberta
  - BC Diabetes, Vancouver, British Columbia
  - LMC Diabetes & Endocrinology Ltd. - Brampton, Brampton, Ontario
  - LMC Diabetes & Endocrinology Ltd. - Thornhill, Concord, Ontario
  - LMC Diabetes & Endocrinology Ltd. - Etobicoke, Etobicoke, Ontario
  - Centre for Studies in Family Medicine, Western Centre for Public Health and Family Medicine, Western University, London, Ontario
  - LMC Diabetes & Endocrinology Ltd. - Toronto, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Québec, Quebec
- Czechia (3):
  - Edumed s.r.o., Jaroměř
  - Nemocnice Pardubickeho kraje, a.s., Nemocnice Pardubice, Pardubice
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (4):
  - Hôpital Jean-Verdier - AP-HP; Service Endocrinologie Diabétologie Nutrition, Bondy
  - CHU Henri Mondor, Créteil
  - CHU de Nantes, Clinique d'Endocrinologie, Nantes
  - Centre Hospitalier de Valenciennes, Valenciennes
- Germany (5):
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder), Brandenburg
  - Herz-und Diabeteszentrum NRW Universitaetsklinik der Ruhr-Universitaet Bochum, Bad Oeynhausen, North Rhine-Westphalia
  - Cardiologicum Pirna und Dresden, Dresden, Saxony
  - Klinische Forschung Berlin GbR, Berlin
  - ZKS - Zentrum Klinische Studien Sudbrandenburg GmbH, Elsterwerda
- Hong Kong (2):
  - Erik Yee Mun George Fung, Shatin
  - Prince of Wales Hospital; Chinese University of Hong Kong; Dept of Medicine and Therapeutics, Shatin
- Poland (9):
  - Centrum Chorob Serca w USK, Wroclaw, Borowska
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok
  - Topolowa MEDICENTER Mrózek & wspólnicy sp.j., Krakow
  - Centrum Twojego Zdrowia, Krakow
  - ETG Lodz, Lodz
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Prywatny Gabinet Lekarski Centrum Medyczne Diabetika, Radom
  - Centrum Medyczne Medyk Stanislaw Mazur Sp. z o.o. SK, Rzeszów
  - 4 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny ZOZ we Wroclawiu, Wroclaw
- Spain (7):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Abente y Lago (Complejo Universitario de la Coruña), A Coruña
  - Hospital de la Santa Creu i Sant Pau Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (5):
  - Ninewells Hospital & Medical School, Dundee
  - CPS Research, Glasgow
  - Glenfield hospital, Leicester
  - Barts and The London School of Medicine & Dentistry, London
  - Wythenshawe Hospital, Manchester

REFERENCES:
- [Derived] Blumer V, Januzzi JL Jr, Liu Y, Butler J, Ezekowitz JA, Perfetti R, Rosenstock J, Del Prato S, Tang WHW, Urbinati A, Zannad F, Lewis GD, Solomon SD, Hedge S, Ibrahim NE, Lam CSP. Sex Differences in Diabetic Cardiomyopathy and Treatment Response to AT-001: Insights From the ARISE-HF Study. JACC Heart Fail. 2025 May 8:102433. doi: 10.1016/j.jchf.2025.02.015. Online ahead of print. PMID 40338768
- [Derived] Siddiqi TJ, Liu Y, Zannad F, Tang WHW, Solomon S, Rosenstock J, Perfetti R, Marwick TH, Lewis GD, Lam CSP, Ibrahim NE, Ezekowitz J, Del Prato S, Butler J, Januzzi JL. Health status in stage B heart failure from diabetic cardiomyopathy baseline results from ARISE-HF. J Diabetes Complications. 2025 Jul;39(7):109059. doi: 10.1016/j.jdiacomp.2025.109059. Epub 2025 Apr 25. PMID 40315802
- [Derived] Tang WHW, Liu Y, Butler J, Del Prato S, Ezekowitz JA, Ibrahim NE, Lam CSP, Marwick TH, Perfetti R, Rosenstock J, Solomon SD, Zannad F, Januzzi JL, Lewis GD. Impaired Exercise Capacity in High-Risk Diabetic Cardiomyopathy: The ARISE-HF Cardiopulmonary Exercise Testing Subanalysis. Circ Heart Fail. 2025 Mar;18(3):e012200. doi: 10.1161/CIRCHEARTFAILURE.124.012200. Epub 2025 Jan 30. PMID 39882614
- [Derived] Marwick TH, Lam C, Liu Y, Del Prato S, Rosenstock J, Butler J, Ezekowitz J, Ibrahim NE, Tang WHW, Zannad F, Perfetti R, Januzzi JL. Echocardiographic phenotypes of diabetic myocardial disorder: evolution over 15 months follow-up in the ARISE-HF trial. Cardiovasc Diabetol. 2025 Jan 13;24(1):16. doi: 10.1186/s12933-024-02554-y. PMID 39806375
- [Derived] Gouda P, Liu Y, Butler J, Del Prato S, Ibrahim NE, Lam CSP, Marwick T, Rosenstock J, Tang W, Zannad F, Januzzi J, Ezekowitz J. Relationship between NT-proBNP, echocardiographic abnormalities and functional status in patients with subclinical siabetic cardiomyopathy. Cardiovasc Diabetol. 2024 Aug 2;23(1):281. doi: 10.1186/s12933-024-02378-w. PMID 39095808
- [Derived] Batista JL, Liu Y, Butler J, Del Prato S, Ezekowitz JA, Lam CSP, Marwick TH, Rosenstock J, Tang WHW, Perfetti R, Urbinati A, Zannad F, Januzzi JL Jr, Ibrahim NE. Racial Differences in Diabetic Cardiomyopathy: The ARISE-HF Trial. J Am Coll Cardiol. 2024 Jul 16;84(3):233-243. doi: 10.1016/j.jacc.2024.04.053. PMID 38986667
- [Derived] Januzzi JL Jr, Butler J, Del Prato S, Ezekowitz JA, Ibrahim NE, Lam CSP, Lewis GD, Marwick TH, Perfetti R, Rosenstock J, Solomon SD, Tang WHW, Zannad F. Randomized Trial of a Selective Aldose Reductase Inhibitor in Patients With Diabetic Cardiomyopathy. J Am Coll Cardiol. 2024 Jul 9;84(2):137-148. doi: 10.1016/j.jacc.2024.03.380. Epub 2024 Apr 8. PMID 38597864
- [Derived] Januzzi JL, Del Prato S, Rosenstock J, Butler J, Ezekowitz J, Ibrahim NE, Lam CSP, Marwick T, Wilson Tang WH, Liu Y, Mohebi R, Urbinati A, Zannad F, Perfetti R. Characterizing diabetic cardiomyopathy: baseline results from the ARISE-HF trial. Cardiovasc Diabetol. 2024 Feb 1;23(1):49. doi: 10.1186/s12933-024-02135-z. PMID 38302936